CLINICAL TRIAL: NCT04085120
Title: Comparison Between Ropivacaine/Dexamethasone and 10% Lignocaine Injection in Distal Glossopharyngeal Nerve Block for Intractable Cancer Pain- A Randomized Trial
Brief Title: Ropivacaine/Dexamethasone and 10% Lignocaine Injection in GPN Block for Intractable Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr.Dinesh Manoharan, Senior Resident, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IEC-402/07.06.2019, RP-34/2019
Record Dates: First submitted 2019-08-11; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Cancer, Oropharynx; Pain, Intractable; Cancer Pain
MeSH Terms: conditions — Oropharyngeal Neoplasms; Pain, Intractable; Cancer Pain | interventions — Ropivacaine; Calcium Dobesilate; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine/dexamethasone group (Experimental): 3ml of 0.75% ropivacaine and 1ml of 4mg/l dexamethasone will be injected.
  Interventions: Procedure: 0.75 % Ropivacaine/ 4mg/mL dexamethasone injection
- 10% lignocaine injection group (Experimental): 4 ml of 10% lignocaine
  Interventions: Procedure: 10% lignocaine injection

INTERVENTIONS:
Procedure: 0.75 % Ropivacaine/ 4mg/mL dexamethasone injection — Distal glossopharyngeal nerve in the neck will be blocked by using 0.75 % Ropivacaine/ 4mg/mL dexamethasone injection
  Arms: Ropivacaine/dexamethasone group
Procedure: 10% lignocaine injection — Distal glossopharyngeal nerve in the neck will be blocked by using 10% lignocaine injection
  Arms: 10% lignocaine injection group

SUMMARY:
The study will compare the efficacy and safety of Ropivacaine/dexamethasone vs 10% lignocaine injection in distal glossopharyngeal nerve block for intractable cancer pain

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven carcinoma of the oropharynx and supraglottic larynx with estimated survival of 3 months or more.
* Pain lasting for at least 2 weeks with an average intensity of 5 or more on an 11-point numeric rating scale (NRS) refractory to a combination strong opioids and NSAIDS

Exclusion Criteria:

1. Local infection or skin ulceration at the puncture site
2. Local anaesthetic allergy
3. Psychiatric illness that affected cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain reduction on the basis of the Numeric rating scale (NRS). | 4 weeks
  Pain reduction on the basis of the Numeric rating scale (NRS). From 0 to 10 (No pain to highest pain)

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI)- short form | 4 weeks
  BPI scores will be used to assess the change in pain before and after treatment. (Likert scale of 0 to 10, where 0 is none to 10 is maximum)
WHO Quality of Life-BREF | 4 weeks
  WHO Quality of Life-BREF scores will be used to assess change in quality of life before and after treatment. (Likert scale of 0 to 5, where 0 is no interference to quality of life and 5 is maximum).
Patient Global Impression of Change (PGIC) | 4 weeeks
  Number of Participants With Treatment Success at the End of Therapy as Measured by the Patient Global Impression of Change (PGIC). A treatment success is defined as Much or Very Much Improved at the Week 4. The PGIC is a 7-point Likert Scale, ranging from very much worse to very much improved
Clinical Global Impression of Change (CGIC) | 4 weeks
  Number of Participants With Treatment Success at the End of Therapy Based on Clinical Global Impression of Change (CGIC) . A treatment success is defined as Much or Very Much Improved at the Week 4. The PGIC is a 7-point Likert Scale, ranging from very much worse to very much improve.
Analgesic requirement and rescue analgesic requirement | 4 weeks
  The number and dose of drugs before and after treatment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Manoharan, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided